CLINICAL TRIAL: NCT01916226
Title: Study 200165, A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Parallel-Group Study to Compare the Efficacy of a 2-Week Treatment With Fluticasone Propionate Nasal Spray Versus Cetirizine in Adult Subjects With Seasonal Allergic Rhinitis (SAR)
Brief Title: A Comparator Study of Fluticasone Propionate Nasal Spray Verses (vs) Cetirizine in the Treatment of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200165
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Rhinitis, Allergic, Perennial and Seasonal
Keywords: cetirizine; seasonal allergic rhinitis; Quality of Life; fluticasone propionate nasal spray
MeSH Terms: conditions — Rhinitis; Rhinitis, Allergic, Seasonal | interventions — Cetirizine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- FPNS arm (Experimental): Subject will receive two sprays (200 mcg per day)of FP into each nostril once daily (OD) every morning for 14 days
  Interventions: Drug: FPNS
- FPNS Placebo arm (Placebo Comparator): Subject will receive two sprays of FP placebo into each nostril OD every morning for 14 days
  Interventions: Drug: FPNS Placebo
- Cetirizine arm (Experimental): Subject will receive Cetirizine capsule by mouth OD in the morning for 14 days
  Interventions: Drug: Cetirizine
- Cetirizine Placebo arm (Placebo Comparator): Subject will receive Cetirizine Placebo capsule by mouth OD in the morning for 14 days
  Interventions: Drug: Cetirizine Placebo

INTERVENTIONS:
Drug: FPNS — Bottled, 16 gm net fill weight for 120 metered sprays with unit dose strength of 50 mcg per spray.
  Arms: FPNS arm
Drug: FPNS Placebo — Bottled placebo nasal spray (vehicle for Fluticasone propionate aqueous nasal spray), 16 gm net fill weight for 120 metered sprays.
  Arms: FPNS Placebo arm
Drug: Cetirizine — Over-encapsulated Cetirizine tablet with unit dose strength of 10 mg in High Density Poly Ethylene Bottles (20 count per bottle).
  Arms: Cetirizine arm
Drug: Cetirizine Placebo — Over-encapsulated Cetirizine matching tablet High Density Poly Ethylene Bottles (20 count per bottle).
  Arms: Cetirizine Placebo arm

SUMMARY:
This phase IV investigational trial is being conducted to evaluate the efficacy of a 2-week treatment of fluticasone propionate nasal spray (FPNS) vs. cetirizine on allergic nasal and ocular symptoms and quality of life in adult subjects with SAR. It is hypothesized that FPNS provides greater nasal symptom relief than cetirizine. The primary measure used to test this hypothesis is the change from baseline over two weeks in reflective total nasal symptom score (rTNSS) compared between FPNS and cetirizine. Approximately 648 subjects will be randomized into a 1:1:1:1 ratio of treatment allocation across approximately twenty-five to thirty-five sites in the US during the 2013 fall allergy season. All subjects will be outpatients. The total duration of study will be approximately 21 days including 7 days of screening period, and 14 days of treatment period.

ELIGIBILITY:
Inclusion Criteria

* Informed consent: Subject must give their signed and dated written informed consent to participate. Subject must understand and be willing, able, and likely to comply with study procedures and restrictions. Subject must be able to read, comprehend, and record information in English.
* Subject is treatable on an outpatient basis.
* Age: >=18 years of age at Visit 1.
* Gender: Male or eligible female subjects. A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g., age appropriate, history of vasomotor symptoms. OR Childbearing potential with a negative pregnancy test at screening and agreeable to using one of the acceptable contraceptive methods consistently and correctly (i.e., in accordance with the approved product label and the instructions of the physician for the duration of the study). An eligible female is also not lactating nor planning on becoming pregnant during the study.
* Diagnosis of SAR, defined as documented clinical history or physician verification of subject reported historical SAR during each of the last two fall allergy seasons and a positive skin prick test (wheal >=3 millimeter [mm] larger than the negative control) to a prevalent local fall allergen within 12 months prior to Visit 1 or at Visit 1.
* Adequate exposure to local fall pollen: Subject resides within a geographical region where exposure to the local fall pollen to which they are sensitized is expected to be moderate or greater during the study period. Subject does not plan to travel outside the geographical region where exposure to local fall pollen to which they are sensitized is expected to be moderate or greater for more than 48 hours during the study period.

At Visit 2, the subject must meet the following criteria

* Eligible subjects will need to have moderate to severe SAR symptoms, defined as a morning rTNSS of >=7 on at least four of the last seven days leading up to randomization. This includes the AM assessment on the morning of the randomization visit at Visit 2.
* Subjects should demonstrate at least a 70% compliance rate with both their placebo run-in study medications and their e-diary completion prior to randomization. This period includes the day of Visit 1 until the day before randomization at Visit 2.
* Subjects should have no significant change in medical condition(s) that would have been exclusionary at Visit 1.
* Subjects should not have used any prohibited medications that are detailed in the inclusion/exclusion criteria (including prohibited allergy medications).
* Subjects should not have travelled outside the local pollen region for more than 48 hours during the run-in period.

Exclusion Criteria

* Significant concomitant medical conditions, defined as but not limited to:

Historical or current evidence of a clinically significant uncontrolled disease of any body system (e.g., tuberculosis, psychological disorders, eczema, uncontrolled asthma). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or which would confound the interpretation of the study results if the disease/condition exacerbated during the study.

A severe physical obstruction of the nose (e.g., deviated septum or nasal polyp) or nasal septal perforation that could affect the deposition of intranasal study drug.

Nasal (e.g., nasal septum), ocular, or throat injury, or surgery to these areas in the last 3 months.

Rhinitis medicamentosa. Bacterial or viral infection (e.g., common cold) of the eyes or upper respiratory tract within two weeks of Visit 1 or during the screening period.

Documented evidence of acute or significant chronic sinusitis, as determined by the individual investigator.

Current or history of glaucoma and/or cataracts or ocular herpes simplex. Physical impairment that would affect subject's ability to safely and fully participate in the study.

Clinical evidence of a Candida infection of the nose. History of psychiatric disease, intellectual deficiency, poor motivation, substance abuse (including drug and alcohol) or other conditions that will limit the validity of informed consent or that would confound the interpretation of the study results.

History of adrenal insufficiency.

* Use of corticosteroids, defined as: Intranasal corticosteroid within four weeks prior to Visit 1 and during the treatment period. Inhaled, oral, intramuscular, intravenous, ocular, and/or dermatological corticosteroid (with the exception of hydrocortisone cream/ointment, 1% or less) within eight weeks prior to Visit 1 and during the treatment period.
* Use of allergy medications, within a timeframe relative to Visit 1, that would prevent the medication from being eliminated and/or have an effect. Exclusionary timeframes relative to Visit 1 for five common allergy treatments are noted below Intranasal cromolyn (<=2 weeks from Visit 1). Intranasal or systemic decongestants (<=3 days from Visit 1). Intranasal or systemic (other than oral) antihistamines (<=3 days from Visit 1).

Leukotriene modifiers (<=3 days from Visit 1). Oral antihistamines (<=2 days from Visit 1). Allergy medications, other than study supplied medications, are not allowed during the study.

* Use of other medications that may affect allergic rhinitis or its symptoms, e.g., use of any ocular antihistamines, artificial tears, eyewashes/nasal irrigation solutions, homeopathic preparations, lubricants, sympathomimetic or vasoconstrictor preparations during the screening and treatment periods
* Use of any medications (prescription or non-prescription) or alcohol to induce sleep 48-hours prior to Visit 1 and during the treatment period.
* Use of other intranasally administered medications (e.g., calcitonin), including herbals and homeopathics during the run-in (Visit 1 - Visit 2) and treatment period.
* Use of immunosuppressive medications within 8 weeks prior to screening and during the treatment period.
* Use of any medications that significantly inhibit the cytochrome P450 subfamily enzyme CYP3A4 (e.g., ritonavir, ketoconazole) during the run-in (Visit 1 - Visit 2) and treatment period.
* Known hypersensitivity to corticosteroids or any excipients present in the nasal spray.
* Known hypersensitivity to cetirizine or any excipients in the tablet.
* Recent exposure to an investigational study drug or device within 30 days of Visit 1.
* Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or immediate family members of the aforementioned are excluded from participating in this study.
* Chickenpox or measles during the last 3 weeks prior to screening and is non-immune.
* Immunotherapy is exclusionary unless the immunotherapy was initiated >=30 days from Visit 1 and if the dose has remained fixed over the 30 days prior to Visit 1, and the dose will remain fixed for the duration of the study.
* Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years which in the opinion of the investigator could interfere with the subject's proper completion of the protocol requirement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2013-08-01; Primary Completion 2013-10-01 (Actual); Study Completion 2013-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- United States (30):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Kerrville, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Greenfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Ford LB, Matz J, Hankinson T, Prillaman B, Georges G. A comparison of fluticasone propionate nasal spray and cetirizine in ragweed fall seasonal allergic rhinitis. Allergy Asthma Proc. 2015 Jul-Aug;36(4):313-9. doi: 10.2500/aap.2015.36.3860. PMID 26108088
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 200165 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200165 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200165 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200165 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200165 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200165 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200165 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In anticipation of a 5% to 8% dropout rate, this study planned enrolment of 156 participants per treatment group in order to target 144 participants per treatment group, who would provide a full 2 weeks' worth of data.
Pre-assignment Details: A total of 978 participants were screened for this study. Of these, 73 were pre-screen failures and 223 were screening/run-in failures. A total of 682 participants were randomized (1:1:1:1 ratio) to receive study treatment.
Groups:
- FPNS 200 μg: Participants self-administered fluticasone propionate nasal spray (FPNS) 200 micrograms (µg) per day as two sprays in each nostril (50 μg per spray) once daily in the morning (AM) for 2 weeks.
- Cetirizine 10 mg: Participants self-administered a 10 milligram (mg) cetrizine capsule once daily in the AM for 2 weeks.
- FPNS Matching Placebo: Participants self-administered matching placebo to FPNS as two sprays in each nostril (50 µg per spray) once daily in the AM for 2 weeks.
- Cetirizine Matching Placebo: Participants self-administered matching placebo to cetrizine capsule once daily in the AM for 2 weeks.
Period: Overall Study
Arm/Group | FPNS 200 μg | Cetirizine 10 mg | FPNS Matching Placebo | Cetirizine Matching Placebo
Started | 170 | 170 | 171 | 171
Completed | 169 | 169 | 168 | 167
Not Completed | 1 | 1 | 3 | 4
Not completed — Adverse Event | 1 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- FPNS 200 μg: Participants self-administered FPNS 200 µg per day as two sprays in each nostril (50 μg per spray) once daily in the AM for 2 weeks.
- Cetirizine 10 mg: Participants self-administered a 10 mg cetrizine capsule once daily in the AM for 2 weeks.
- Total: Total of all reporting groups
Arm/Group | FPNS 200 μg | Cetirizine 10 mg | FPNS Matching Placebo | Cetirizine Matching Placebo | Total
Number analyzed (Participants) | 170 | 170 | 171 | 171 | 682
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.1 (10.66) | 39.2 (11.41) | 41.3 (11.29) | 40.4 (11.84) | 40.3 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 113 | 110 | 109 | 428
  Male | 74 | 57 | 61 | 62 | 254
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 34 | 20 | 31 | 35 | 120
  American Indian or Alaska Native | 1 | 0 | 1 | 1 | 3
  Asian - Central/South Asian Heritage | 2 | 2 | 5 | 3 | 12
  Asian-East Asian Heritage | 1 | 0 | 1 | 0 | 2
  Asian - South East Asian Heritage | 2 | 0 | 1 | 2 | 5
  White - Arabic/North African Heritage | 1 | 0 | 1 | 1 | 3
  White - White/Caucasian/European Heritage | 129 | 142 | 128 | 127 | 526
  Mixed Race | 0 | 6 | 3 | 1 | 10
  Not Captured by Study Site | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (CFB) in the Individual AM Reflective Total Nasal Symptom Scores (rTNSS) Over the Entire Treatment Period
Description: The rTNSS score is the sum of the four individual symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing. Each symptom is scored on a scale ranging from 0 to 3; the rTNSS ranges from 0 (none) to 12 (severe). Each individual symptom was evaluated using a scale of 0 (none), 1 (mild), 2 (moderate), or 3 (severe). The reflective assessment of the TNSS scores the four nasal symptoms over the previous 24 hours. The participants themselves scored nasal symptoms in an e-diary. Baseline is defined as the arithmetic average of the rTNSS recorded on the morning of randomization and on each of the six preceding days. A participant may have had as few as 4 days' worth of data contributing to the Baseline average. The 2-week symptom score was defined as the average of the values recorded on the day after randomization and the following 13 days. Change from Baseline was thus calculated as the 2-week average minus the Baseline value.
Time Frame: Baseline through the entire treatment period (2 weeks)
Population: Intent-to-Treat (ITT) Population: all participants who were randomized and received at least one dose of study medication. Change from Baseline was analyzed for only those participants who were available for assessment at Baseline and at Weeks 1 and 2.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | FPNS 200 μg | Cetirizine 10 mg | FPNS Matching Placebo | Cetirizine Matching Placebo
Number analyzed (Participants) | 169 | 169 | 171 | 171
Scores on a scale | -2.2 (0.19) | -1.9 (0.18) | -1.5 (0.18) | -0.9 (0.16)
Statistical Analysis 1: Comparison: FPNS 200 μg vs Cetirizine 10 mg; Test type: Superiority or Other; p = 0.278, ANCOVA — Estimating the standard deviation of CFB in rTNSS over 2 weeks to be approximately 2.6, a two-sample t-test with α=0.05 suggests that a sample size of 144 participants per arm would provide 90% power to show a difference of 1.0 between treatments; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-0.7 to 0.2], Standard Error of Mean -0.3

2. Secondary Outcome: Mean Change From Baseline in the Individual AM Reflective Nasal Symptom Scores for Rhinorrhea, Nasal Congestion, Nasal Itching, and Sneezing Over the Entire Treatment Period
Description: Each individual symptom was evaluated using a scale of 0 (none), 1 (mild), 2 (moderate), or 3 (severe).The reflective assessment scores the four nasal symptoms over the previous 24 hours. The participants themselves scored nasal symptoms in an e-diary. Baseline is defined as the arithmetic average of the individual AM reflective nasal symptom scores recorded on the morning of randomization and on each of the six preceding days. A participant may have had as few as 4 days' worth of data contributing to the Baseline average. The 2-week symptom score was defined as the average of the values recorded on the day after randomization and the following 13 days. Change from Baseline was thus calculated as the 2-week average minus the Baseline value.
Time Frame: Baseline through the entire treatment period (2 weeks)
Population: ITT Population. Change from Baseline was analyzed for only those participants who were available for assessment at Baseline and at Weeks 1 and 2.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | FPNS 200 μg | Cetirizine 10 mg | FPNS Matching Placebo | Cetirizine Matching Placebo
Number analyzed (Participants) | 169 | 169 | 171 | 171
Scores on a scale
  Nasal congestion | -0.5 (0.05) | -0.4 (0.04) | -0.3 (0.05) | -0.2 (0.04)
  Nasal itching | -0.6 (0.05) | -0.5 (0.05) | -0.4 (0.05) | -0.2 (0.04)
  Runny nose | -0.5 (0.05) | -0.4 (0.05) | -0.4 (0.05) | -0.3 (0.05)
  Sneezing | -0.6 (0.05) | -0.6 (0.05) | -0.4 (0.05) | -0.2 (0.05)

3. Secondary Outcome: Mean Change From Baseline in the Nocturnal Rhinoconjunctivitis Quality of Life Questionnaire (NRQLQ) Overall Score at Visit 3/Early Withdrawal.
Description: The NRQLQ is a 16-item, validated, self-administered, disease (allergic rhinitis)-specific quality of life instrument that measures the functional problems most troublesome to participants with nocturnal allergy symptoms over a one-week interval. Each question is scored on a 7-point scale from 0 (not troubled) to 6 (extremely troubled). Items are grouped into four domains: sleep problems (4 items), sleep time problems (5 items), symptoms on waking in the morning (4 items), and practical problems (3 items). An overall score was calculated from the individual item scores. All items are weighted equally. A mean score is calculated across all items within each domain. The overall score is the mean across all items and ranges from 0 (not troubled) to 6 (extremely troubled). Higher scores reflect a lower quality of life. Change from Baseline was calculated as the 2-week average minus the Baseline value.
Time Frame: Baseline and Visit 3 (Study Day 14 +/- 2 days)/Early Withdrawal
Population: ITT Population
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | FPNS 200 μg | Cetirizine 10 mg | FPNS Matching Placebo | Cetirizine Matching Placebo
Number analyzed (Participants) | 170 | 170 | 171 | 171
Scores on a scale | -1.0 (0.10) | -0.6 (0.09) | -0.8 (0.10) | -0.5 (0.08)

4. Secondary Outcome: Mean Change From Baseline in the AM Pre-dose Instantaneous Total Nasal Symptom Score (iTNSS) Over the Entire Treatment Period
Description: The iTNSS score is the sum of the four individual symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing. Each symptom is scored on a scale ranging from 0 to 3; the iTNSS ranges from 0 (none) to 12 (severe). The symptoms were evaluated using a scale of 0 (none), 1 (mild), 2 (moderate), or 3 (severe). The instantaneous assessment of the TNSS scores the four nasal symptoms at the time of the assessment, or at that "instant." The participants themselves scored nasal symptoms in an e-diary once each morning prior to administering study drug. Baseline is defined as the arithmetic average of the iTNSS recorded on the morning of randomization and on each of the six preceding days. A participant may have had as few as 4 days' worth of data contributing to the Baseline average. The 2-week symptom score was defined as the average of the values recorded on the day after randomization and the following 13 days.
Time Frame: Baseline through the entire treatment period (2 weeks)
Population: ITT Population. Change from Baseline was analyzed for only those participants who were available for assessment at Baseline and at Weeks 1 and 2. Change from Baseline was calculated as the 2-week average minus the Baseline value.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | FPNS 200 μg | Cetirizine 10 mg | FPNS Matching Placebo | Cetirizine Matching Placebo
Number analyzed (Participants) | 169 | 169 | 171 | 171
Scores on a scale | -1.9 (0.18) | -1.3 (0.17) | -1.2 (0.18) | -0.6 (0.15)

5. Secondary Outcome: Mean Change From Baseline in the AM Pre-dose Reflective Total Ocular Symptom Score (rTOSS) Over the Entire Treatment Period
Description: The rTOSS is an eye assessment that comprises the sum of the three symptom scores for tearing/watering, itching/burning, and eye redness. Each symptom is scored on a scale of 0 to 3: 0, none; 1, mild; 2, moderate; 3, severe. The rTOSS ranges from 0 (none) to 9 (severe). The reflective assessment scores the participants' ocular symptoms over the preceding 24 hours. The participants themselves scored ocular symptoms in an e-diary. Baseline arithmetic is defined as the average of the rTNSS recorded on the morning of randomization and on each of the six preceding days. A participant may have had as few as 4 days' worth of data contributing to the Baseline average. The 2-week symptom score was defined as the average of the values recorded on the day after randomization and the following 13 days. Change from Baseline was thus calculated as the 2-week average minus the Baseline value.
Time Frame: Baseline through the entire treatment period (2 weeks)
Population: Ocular Population: all ITT participants with a Baseline rTOSS of 4 or greater
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | FPNS 200 μg | Cetirizine 10 mg | FPNS Matching Placebo | Cetirizine Matching Placebo
Number analyzed (Participants) | 150 | 137 | 152 | 146
Scores on a scale | -1.6 (0.16) | -1.4 (0.16) | -1.2 (0.16) | -0.8 (0.14)

6. Secondary Outcome: Mean Change From Baseline in the AM Pre-dose Instantaneous Total Ocular Symptom Score (iTOSS) Over the Entire Treatment Period
Description: The iTOSS is an eye assessment that comprises the sum of the three symptom scores for tearing/watering, itching/burning, and eye redness. Each symptom is scored on a scale of 0 to 3: 0, none; 1, mild; 2, moderate; 3, severe. The iTOSS ranges from 0 (none) to 9 (severe). The instantaneous assessment scores the participants' ocular symptoms at the time of the assessment, or at that "instant." The participants themselves scored ocular symptoms in an e-diary once each morning prior to administering study drug. Baseline is defined as the arithmetic average of the iTOSS recorded on the morning of randomization and on each of the six preceding days. A participant may have had as few as 4 days' worth of data contributing to the Baseline average. The 2-week symptom score was defined as the average of the values recorded on the day after randomization and the following 13 days. Change from Baseline was thus calculated as the 2-week average minus the Baseline value.
Time Frame: Baseline through the entire treatment period (2 weeks)
Population: Ocular Population
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | FPNS 200 μg | Cetirizine 10 mg | FPNS Matching Placebo | Cetirizine Matching Placebo
Number analyzed (Participants) | 150 | 137 | 152 | 146
Scores on a scale | -1.3 (0.15) | -1.1 (0.14) | -1.1 (0.16) | -0.5 (0.13)

7. Secondary Outcome: Mean Change From Baseline in the Combined Nasal and Ocular Reflective Total Symptom Score (rTSS = rTNSS+rTOSS) Over the Entire Treatment Period
Description: The rTSS is the sum of the rTNSS and the rTOSS. The rTNSS score is the sum of the four individual symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing. Each symptom is scored on a scale ranging from 0 to 3; the rTNSS ranges from 0 (none) to 12 (severe). Each individual symptom was evaluated using a scale of 0 (none), 1 (mild), 2 (moderate), or 3 (severe). The rTOSS assessment is comprised of the sum of the three symptom scores for tearing/watering, itching/burning, and eye redness. Each symptom is scored on a scale of 0 to 3: 0, none; 1, mild; 2, moderate; or 3, severe. The rTOSS ranges from 0 (none) to 9 (severe). The reflective assessment scores participants' symptoms over the previous 24 hours. The participants themselves scored nasal and ocular symptoms in an e-diary. Baseline is defined as the arithmetic average of the rTSS recorded on the morning of randomization and on each of the six preceding days.
Time Frame: Baseline through the entire treatment period (2 weeks)
Population: Ocular Population. Change from Baseline was calculated as the 2-week average minus the Baseline value.n
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | FPNS 200 μg | Cetirizine 10 mg | FPNS Matching Placebo | Cetirizine Matching Placebo
Number analyzed (Participants) | 150 | 137 | 152 | 146
Scores on a scale | -3.9 (0.34) | -3.4 (0.34) | -2.7 (0.34) | -1.7 (0.30)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment until the End-of-Study visit (up to Day 14).
Description: SAEs and non-serious AEs are reported for the Intent-to-Treat Population, comprised of all participants who were randomized and received at least one dose of study medication.
Arm/Group | FPNS 200 μg | Cetirizine 10 mg | FPNS Matching Placebo | Cetirizine Matching Placebo
Serious Adverse Events (participants affected / at risk) | 0/170 | 0/170 | 0/171 | 0/171
Other Adverse Events (participants affected / at risk) | 10/170 | 13/170 | 10/171 | 10/171
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FPNS 200 μg (N=170) | Cetirizine 10 mg (N=170) | FPNS Matching Placebo (N=171) | Cetirizine Matching Placebo (N=171)
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 3 | 2 | 3
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.